CLINICAL TRIAL: NCT00077155
Title: A Phase I Study Of Continuous Infusion EMD 121974 In Patients With Solid Tumors
Brief Title: Cilengitide (EMD 121974) in Treating Patients With Advanced Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02569; UCCRC-12774A; CDR0000349535 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-02-10; First posted 2004-02-11 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: AIDS-related Peripheral/Systemic Lymphoma; AIDS-related Primary CNS Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Splenic Marginal Zone Lymphoma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Mycosis Fungoides/Sezary Syndrome; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Mycosis Fungoides/Sezary Syndrome; Stage IV Small Lymphocytic Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cilengitide

ARMS (1):
- Treatment (cilengitide) (Experimental): Patients receive cilengitide (EMD 121974) IV continuously on weeks 1-4. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of EMD 121974 until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  Interventions: Drug: cilengitide

INTERVENTIONS:
Drug: cilengitide
  Other Names: EMD 121974

SUMMARY:
This phase I trial is studying the side effects and best dose of EMD 121974 in treating patients with solid tumors or lymphoma. Cilengitide (EMD 121974) may stop the growth of cancer cells by stopping blood flow to the cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the dose-limiting toxicity, maximum feasible dose, and recommended phase II dose of cilengitide (EMD 121974) in patients with advanced solid tumors or lymphoma.

II. Determine the safety and tolerability of this drug in these patients.

SECONDARY OBJECTIVES:

I. Determine the pharmacokinetics of this drug in these patients. II. Determine the antineoplastic activity of this drug in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive cilengitide (EMD 121974) IV continuously on weeks 1-4. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of EMD 121974 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor or lymphoma
* Refractory to standard therapy or no standard therapy exists
* Measurable or evaluable disease
* No active brain metastases

  * Previously treated brain metastases allowed provided the patient is not currently receiving corticosteroids
  * Primary brain neoplasms allowed, regardless of corticosteroid use
* Performance status - Karnofsky 70-100%
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* No life-threatening bleeding diathesis within the past 6 months
* Bilirubin normal (unless due to Gilbert's syndrome)
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No prior proven gastric or duodenal ulcer
* No clinically significant gastrointestinal blood loss within the past 6 weeks
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior CNS hemorrhage
* No psychiatric illness or social situation that would preclude study compliance
* No other concurrent uncontrolled illness
* No ongoing or active infection
* No prior cilengitide (EMD 121974)
* No other concurrent biologic therapy
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No concurrent chemotherapy
* See Disease Characteristics
* More than 4 weeks since prior radiotherapy and recovered
* No concurrent palliative radiotherapy
* No other concurrent anticancer agents or therapies intended to treat the malignancy
* No other concurrent investigational agents
* No concurrent anticoagulation therapy that increases INR or aPTT above the normal range

  * Line prophylaxis allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2003-12; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Maximum feasible dose defined as the highest dose studied for which the incidence of DLT is less than 33% or the highest safe dose in our study, limited to a maximum MFD dose of 40 mg/hr | 4 weeks

SECONDARY OUTCOMES:
Pharmacokinetics of EMD 121974 | Up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Samir Undevia, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States